CLINICAL TRIAL: NCT01416649
Title: Impact of Exenatide on Sleep Duration and Quality in Type 2 Diabetes
Brief Title: Impact of Exenatide on Sleep Duration
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-051-A
Record Dates: First submitted 2011-08-11; First posted 2011-08-15 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Exenatide — Exenatide is started for the treatment of type 2 diabetes as determined by the patients regular physician. The dose will be 5-10 micrograms twice daily which is the standard dose. The medication is given by self-administered subcutaneous injection. The medication may continue for the treatment of the type 2 diabetes after the study is completed after 3 months.
  Other Names: The brand name of exenatide is Byetta.

SUMMARY:
This study investigates the effect of exenatide, a FDA approved medication for the treatment of type 2 diabetes on sleep duration and quality. Individuals with type 2 diabetes will be studied before and during treatment with Exenatide.

Enrolled individuals will be asked to come to the University of Chicago for 3-4 outpatient visits over the course of 3-4 months.

ELIGIBILITY:
Inclusion Criteria:

Patients taking diabetes medications other then insulin will be included, but changes to their medications may be made as deemed necessary by their physician. Patients on stable medications for chronic and co-morbid conditions (high blood pressure, high cholesterol, etc) will be eligible

Exclusion Criteria:

Patients with moderate or severe kidney disease and history of pancreatitis or patients on insulin will be excluded, as Exenatide use is contraindicated or risky in these conditions.

Patients with unstable cardiac, neurological or psychiatric disease and women who are pregnant or trying to get pregnant will be excluded. Patients who have severe COPD, severe neuropathy or chronic pain, which could impair sleep, will be excluded. Shift workers will be also excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience Sample
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Sleep duration and sleep efficiency | at the end of 3 months of treatment with the medication
  Sleep duration and efficiency will be measured using an activity monitor worn on the wrist.

CONTACTS AND LOCATIONS:
Overall Officials: Silvana Pannain, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States